CLINICAL TRIAL: NCT04763122
Title: Decline in Radioiodine Use But Not Total Thyroidectomy in Thyroid Cancer Patients Treated in United Arab Emirates- A Retrospective Study
Brief Title: Thyroid Cancer in United Arab Emirates
Status: Completed | Type: Observational
Sponsor: Tawam Hospital (Other)
Responsible Party: Principal Investigator, Khaled M Aldahmani, Consultant Endocrinologist, Tawam Hospital
Other Study IDs: SA/AJ/562
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Thyroid; Cancer
Keywords: Malignancy; Radioactive iodine; total thyroidectomy; Thyroid Cancer
MeSH Terms: conditions — Thyroid Diseases; Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid Cancer Cases
  Interventions: Other: not applicable as it is a retrospective study

INTERVENTIONS:
Other: not applicable as it is a retrospective study — It is a retrospective study

SUMMARY:
The main objective of the study is to assess the trend of clinicopathological features and treatment modalities in patients with thyroid cancer in the largest oncology center in the United Arab Emirates (UAE).

DETAILED DESCRIPTION:
The aim of this study is to assess the trend of clinicopathological features and treatment modalities in patients with thyroid cancer (TC) in the largest oncology center in the United Arab Emirates (UAE).

This study was conducted in Tawam hospital (TWM), which provides tertiary care services to patients in the UAE. It is the only center delivering radioactive iodine (RAI) therapy and radiotherapy in Al Ain city. Most TC patients are followed in designated TC clinics within the endocrinology division or less commonly through other clinics (surgery, radiation, or medical oncology). The hospital runs monthly multidisciplinary team-based discussions on patients with TC, wherein decisions regarding RAI treatment and dose selection are determined jointly by nuclear medicine physicians and endocrinologists.

We retrospectively evaluated all patients with TC presenting to TWM during the period of September 2008 and December 2018. The beginning of data collection (September 2008) reflects the inception time of electronic medical records (EMRs) use in the hospital. Cases of TC were extracted from the EMRs using the International Classification of Disease 9 & 10 codes (193 & c73). Other variables were demographic information, year of diagnosis, type of TC, histopathological subtype, lymph node (LN) involvement, type of thyroid surgery, use of RAI treatment, and radiation therapy. The extent of surgery, the exact details of histopathology, and the RAI dose were retrieved from the respective specialty reports. Tumor staging was reported according to the 8th edition of the American joint committee on cancer (AJCC)/TNM staging system [16]. Those with incorrect pathological diagnosis, incomplete data, or noninvasive follicular type PTC were excluded.

The data were extracted using Microsoft Excel 2015 and imported into Stata 16.0 for statistical analysis. Continuous variables were described using means and standard deviations (±SD). Categorical variables were described as frequency distributions. Variables of clinical features and management were cross tabulated with the year of diagnosis and exact logistic and ordinal logistic regressions were performed to analyze the annual trend in features and management of TC as appropriate. The results of relative trend were reported as odds ratio (OR) with an overall ptrend. The OR=1 indicated no change over years, OR <1 indicated a decline, while OR >1 indicated an increase over years. Simple and multiple logistic regression analysis were performed to assess the unadjusted and adjusted association of management of TC (RAI, surgical management) with age, gender, nationality, year of diagnosis, tumor subtype, and other co-variates. The results of simple and multiple logistic regression were reported as odd ratios (OR) and adjusted odds ratios (AOR) respectively with their corresponding 95% confidence intervals (CI) and p-values.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Thyroid Cancer presenting to Tawam Hospital during the period of September 2008 and December 2018.

Exclusion Criteria:

* Patients with inadequate data, noninvasive follicular type PTC and incorrect pathological diagnosis,

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Thyroid Cancer presenting to Tawam Hospital during the period of September 2008 and December 2018. Those with incorrect pathological diagnosis, incomplete data, or noninvasive follicular type PTC were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 762 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Clinicopathological features | September 2008- December 2018
  Assess clinicopathological features of thyroid cancer patients
Extent of surgery | September 2008- December 2018
  Assess extent of surgery in thyroid cancer patients and changes over time
Use of RAI | September 2008- December 2018
  Evaluate the use of RAI in thyroid cancer patients and assess predictors of RAI Rx

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT04763122/Prot_SAP_000.pdf